CLINICAL TRIAL: NCT00082238
Title: Increased Gluconeogenesis is One Cause of CFRD
Brief Title: Increased Gluconeogenesis is One Cause of Cystic Fibrosis Related Diabetes (CFRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 58603DK (completed); R01DK058603 (NIH)
Record Dates: First submitted 2004-05-03; First posted 2004-05-05 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis; Diabetes Mellitus
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cystic fibrosis (CF) (Experimental)
  Interventions: Other: Stable isotopes
- Healthy volunteers (Active Comparator)
  Interventions: Other: Stable isotopes

INTERVENTIONS:
Other: Stable isotopes — Stable isotopes were used to quantify gluconeogenesis GNG, hepatic glucose production (HGP), and protein breakdown.

SUMMARY:
People with CF have a high incidence of diabetes, called CFRD. CFRD is an important cause of worsened morbidity and mortality, thus understanding the pathophysiology underlying its development is imperative. Insulin deficiency has been well recognized as one cause of CFRD; however the clinical presentation and studies of pathogenesis indicate that the etiology is more complex. There is strong evidence that normal metabolism of carbohydrate, protein and fat is altered in CF. We believe that the inflammatory response to chronic underlying lung disease is responsible for insulin resistance and alters substrate metabolism, and that these changes, in addition to insulin deficiency cause CFRD. Our global hypothesis is that hyperglycemia is caused, in part, by high rates of gluconeogenesis resulting from excessive amino acid substrate availability caused by cytokine-mediated protein catabolism. We further hypothesize that inflammation alters normal fatty acid metabolism leading to lipogenesis, an energy wasteful pathway. We will recruit 24 adult CF subjects and 10 controls (similar in distribution in lean tissue mass, age and gender) and will categorize them according to glucose tolerance (OGTT), as well as insulin secretion and insulin sensitivity using the Tolbutamide-stimulated IVGTT and the Minimal Model. Clinical status will be characterized by measuring pulmonary function and modified NIH scores, in addition to measuring levels of circulating cytokines. Gluconeogenesis (GNG) will be quantified by measuring the incorporation 2H into the 2nd, 5th and 6th carbons of glucose. Amino acid turnover rates will be measured using stable isotopes of lactate and alanine and whole body protein turnover (WBPT) will be measured using [1-13C]leucine and [15N2]urea. Fat metabolism will be evaluated by measuring ketone body turnover using stable isotopes, and by quantifying lipogenesis using the isotopomer equilibration method. Key enzymes of fatty acid metabolism will also be measured. We will utilize indirect calorimetry to measure resting energy expenditure. Subjects will be recruited from the CF centers at the University of Texas- Southwestern and the South Central CF Consortium.

DETAILED DESCRIPTION:
People with CF have a high incidence of diabetes, called CFRD. CFRD is an important cause of worsened morbidity and mortality, thus understanding the pathophysiology underlying its development is imperative. Insulin deficiency has been well recognized as one cause of CFRD; however the clinical presentation and studies of pathogenesis indicate that the etiology is more complex. There is strong evidence that normal metabolism of carbohydrate, protein and fat is altered in CF. We believe that the inflammatory response to chronic underlying lung disease is responsible for insulin resistance and alters substrate metabolism, and that these changes, in addition to insulin deficiency cause CFRD. Our global hypothesis is that hyperglycemia is caused, in part, by high rates of gluconeogenesis resulting from excessive amino acid substrate availability caused by cytokine-mediated protein catabolism. We further hypothesize that inflammation alters normal fatty acid metabolism leading to lipogenesis, an energy wasteful pathway. We will recruit 24 adult CF subjects and 10 controls (similar in distribution in lean tissue mass, age and gender) and will categorize them according to glucose tolerance (OGTT), as well as insulin secretion and insulin sensitivity using the Tolbutamide-stimulated IVGTT and the Minimal Model. Clinical status will be characterized by measuring pulmonary function and modified NIH scores, in addition to measuring levels of circulating cytokines. Gluconeogenesis (GNG) will be quantified by measuring the incorporation 2H into the 2nd, 5th and 6th carbons of glucose. Amino acid turnover rates will be measured using stable isotopes of lactate and alanine and whole body protein turnover (WBPT) will be measured using [1-13C]leucine and [15N2]urea. Fat metabolism will be evaluated by measuring ketone body turnover using stable isotopes, and by quantifying lipogenesis using the isotopomer equilibration method. Key enzymes of fatty acid metabolism will also be measured. We will utilize indirect calorimetry to measure resting energy expenditure. Subjects will be recruited from the CF centers at the University of Texas- Southwestern and the South Central CF Consortium.

Our proposal is intended to better describe the unique metabolism of people with CF, and to provide a comprehensive evaluation of pathophysiologic changes which contribute to the development of CFRD and to wasting; and are part of the applicant's long-range goal which is to identify the underlying causes of CF related diabetes and catabolism so that disease-specific therapies can be developed. We fully expect that the proposed studies will provide new and important information.

ELIGIBILITY:
cystic fibrosis with any type of glucose tolerance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

REFERENCES:
- [Result] Hardin DS, Ahn C, Rice J, Rice M, Rosenblatt R. Elevated gluconeogenesis and lack of suppression by insulin contribute to cystic fibrosis-related diabetes. J Investig Med. 2008 Mar;56(3):567-73. doi: 10.2310/JIM.0b013e3181671788. PMID 18418124